CLINICAL TRIAL: NCT04933058
Title: Opioid Based Analgesia vs Non-opioid Analgesia for Oocyte Retrieval Procedure - a Randomized Clinical Trial
Brief Title: Opioid Based Analgesia vs Non-opioid Analgesia for Oocyte Retrieval Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1025-20-TLV
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Women Undergoing Oocyte Retrieval Procedures
MeSH Terms: interventions — Acetaminophen; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free anesthesia (Experimental): 1. IV propofol 1-1.5 mg/kg
  2. IV acetaminophen 1000mg
  3. IV dipyrone 1000mg
  4. IV lidocaine 1mg/kg
  5. IV dexacort 4mg
  6. PR diclofenac 50 mg
  Interventions: Drug: IV acetaminophen
- Opioid-supplemented anesthesia (Active Comparator): 1. IV propofol 1-1.5 mg/kg
  2. IV fentanyl 1.5 mcg/kg
  3. IV dipyrone 1000mg
  4. IV lidocaine 1mg/kg
  5. IV dexacort 4mg
  6. PR diclofenac 50 mg
  Interventions: Drug: IV fentanyl

INTERVENTIONS:
Drug: IV acetaminophen — Pain management
  Arms: Opioid-free anesthesia
Drug: IV fentanyl — Pain management
  Arms: Opioid-supplemented anesthesia

SUMMARY:
It is unclear whether routine addition of opioids for analgesia during minor gynecological procedures is beneficial. In this single-center randomized single-blinded trial, the investigators aim to test the primary hypothesis that opioid-sparing anesthesia regimen including intravenous acetaminophen is non-inferior to a similar anesthesia regimen containing fentanyl in providing postoperative analgesia in women recovering from oocyte retrieval procedures for in vitro fertilization. The investigators also aim to assess the difference in incidence of patient-reported opioid related adverse-effects between the two groups, time to discharge from the post-anesthesia care unit and postoperative rescue analgesia requirements. If we demonstrate no clinically important difference between the two interventions, clinicians may be able to substantially reduce the amount of opioids administered to patients undergoing minor ambulatory procedures, and potentially decrease the associated opioid related adverse effects.

DETAILED DESCRIPTION:
Study Overview The investigators propose a single-center randomized single-blinded clinical trial in which healthy women undergoing oocyte retrieval procedures under general anesthesia will be randomized to receive either 1.5mcg/kg fentanyl or IV acetaminophen as part of multimodal analgesia. The investigators will evaluate the effects of an opioid-free anesthesia on pain scores, analgesic medication consumption during the initial two postoperative hours, and time to discharge from PACU, compared to an opioid-containing anesthesia.The investigators will also compare the prevalence of opioid-related sedation side effect between opioid-free anesthesia and opioid-containing anesthesia.

Setting and Population Inclusion Criteria

1. Written informed consent 2. 18-45 years old 3. American Society of Anesthesiologists (ASA) physical status 1-2 4. Undergoing oocyte retrieval procedures 5. Planned number of oocytes to be retrieved <15 Exclusion Criteria

1. Known allergy to fentanyl, acetaminophen, dipyrone, lidocaine, propofol or NSAIDs.
2. Endometriosis
3. Diagnosis of chronic pain
4. Opioid dependency, defined by consumption of oral morphine equivalent of greater than or equal to 60mg a day for 7 days or longer, for any time period.
5. Weight < 50 kg
6. Cannabis use
7. Major psychiatric disorder - Schizophrenia, bipolar disorder, major depression.
8. Epilepsy disorder under anti-convulsant therapy.
9. Renal insufficiency, defined as creatinine clearance <60 ml/hr
10. Hepatic disease

Withdrawal Criteria

1. Patients are free to withdraw from the study at any time, for any reason.
2. Patients may be withdrawn from the study by a member of the study team or the clinical team, if seems appropriate for patient's safety or well-being. Examples of such events include (but are not limited) to:

   an allergic reaction, analgesic failure per acute pain service judgement and significant patient discomfort.
3. Reason for exclusion will be documented, and patients will be asked to continue follow-up according to the intention-to-treat principle

Protocol

The investigators propose a randomized, single-blinded single-center clinical trial. After confirming eligibility, patients will be approached before the procedure for possible enrollment in the study. After thorough explanation, written informed consent will be obtained. Patients will be randomized in a 1:1 ratio by a web-based software to receive either:

1. Opioid-free anesthesia, including

   1. IV propofol 1-1.5 mg/kg
   2. IV acetaminophen 1000mg
   3. IV dipyrone 1000mg
   4. IV lidocaine 1mg/kg
   5. IV dexacort 4mg
   6. PR diclofenac 50 mg
2. Opioid-supplemented anesthesia, including

   1. IV propofol 1-1.5 mg/kg
   2. IV fentanyl 1.5 mcg/kg
   3. IV dipyrone 1000mg
   4. IV lidocaine 1mg/kg
   5. IV dexacort 4mg
   6. PR diclofenac 50 mg

The anesthesiologist performing the procedure will not be blinded to group allocation, but other research team members and caregivers who evaluate the patients after the procedure will be.

General anesthesia will be induced according to the group allocation as mentioned above. Anesthesia maintenance will be achieved with 50% N2O via a face-mask, and additional doses of 10-20 mg of propofol as needed. Ketamine will not be allowed. Postoperatively, intravenous tramadol 100 mg will be ordered for breakthrough pain as well as intravenous ondansetron 4mg and metoclopramide 10mg for nausea and vomiting. Patients will be followed until home discharge. The rest of postoperative care will be conducted according to standard departmental procedures by nurses and physicians.

Measurements

* Patient characteristics and demographic data including age, weight, body mass index (BMI), tobacco use, prior IVF treatment, history of pain after previous IVF, chronic pain, chronic medication use, and American Society of Anesthesiologists (ASA) physical status will be obtained from the medical record and patient interview.
* Postoperative pain scores will be documented on an 11-point Numerical Rating Scale (NRS) from 0 (no pain) to 10 (worst pain imaginable) at least once every 30 minutes for the initial two postoperative hours.
* Opioid-induced sedation will be captured through the Passero opioid-induced sedation scale (Appendix A) 20 minutes after patient admission to the recovery room.
* Patient satisfaction with the anesthesia will be assessed using Likert scale from 1 to 5 grading "how satisfied are the participant with the pain management they received today?"
* Time of discharge will be captured from the patient's electronic medical record and/or from patient interview.

Sample Size Considerations To test a unilateral non-inferiority hypothesis, assuming a 2.5% significance level, power of 80%, standard deviation of 2 points, a non-inferiority delta of no more than 1.5 points in the 11-point NRS pain scale between the two groups, and assumed pooled variance of 6, we will need a sample size of 42 patients in each group. Accounting for a predicted loss to follow-up of up to 20% of patients, we aim to recruit 100 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. 18-45 years old
3. American Society of Anesthesiologists (ASA) physical status 1-2
4. Undergoing oocyte retrieval procedures
5. Planned number of oocytes to be retrieved <15

Exclusion Criteria:

1. Known allergy to fentanyl, acetaminophen, dipyrone, lidocaine, propofol or NSAIDs.
2. Endometriosis
3. Diagnosis of chronic pain
4. Opioid dependency, defined by consumption of oral morphine equivalent of greater than or equal to 60mg a day for 7 days or longer, for any time period.
5. Weight < 50 kg
6. Cannabis use
7. Major psychiatric disorder - Schizophrenia, bipolar disorder, major depression.
8. Epilepsy disorder under anti-convulsant therapy.
9. Renal insufficiency, defined as creatinine clearance <60 ml/hr
10. Hepatic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
the difference in average pain scores | 1 year
  We will test the difference in average pain scores between the groups in a non-inferiority model. All pain scores obtained during the initial two postoperative hours will be averaged and compared between the groups. The non-inferiority delta will be defined a priori as no worse than 1.5 points in average pain score. Overall alpha will be 0.05. NRS Scale from 0-10, zero is no pain.
the dependent categorical variable of time-to-discharge readiness | 1 year
  The secondary analysis will compare the dependent variable of time-to-discharge from postanesthesia care unit (PACU) readiness at 60 mins (yes/no) between the two study groups and will be reported as number (proportions). We will also record the time from arrival until discharge from PACU reported as the median [interquartile range] time in each group. Overall alpha will be 0.05.

OTHER OUTCOMES:
comparison of the average sedation scores 20 minutes after admission to the recovery room | 1 year
  We will compare average sedation scores 20 minutes after admission to the recovery room between the groups using a two-sided Student's t-test.
  We will also compare the proportion of patients who required rescue analgesics (tramadol) in PACU between the two groups, using the Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Farladansky, MD, Principal Investigator — senior doctor
Locations (1):
- tel aviv SMO, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No